CLINICAL TRIAL: NCT04766619
Title: Generating Recommendations for National Roll-out and Sustainable Use of Prescribing Safety Indicator Based Interventions Using Longitudinal Process Evaluation and a Consolidated Learning Exercise
Brief Title: Process Evaluation of OptimiseRx and PINCER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 17099
Record Dates: First submitted 2021-01-25; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Medication Errors
Keywords: Medication errors; Primary Care; Prescribing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Staff and stakeholders: For the longitudinal process evaluation - staff and stakeholders who have had direct contact or involvement with and have an understanding of OptmiseRx and/or PINCER will be invited to take part in an interview or focus group, an observation and/or complete a questionnaire. For the consolidated learning exercise - those who are in a position to influence the wider adoption of these interventions will be invited to take part in an interview or development workshop.
- Patients: Patients registered with a practice who have attended a consultation (or other related activity) for the PINCER intervention OR selected by their clinical care team OR attached to a patient group within a Clinical Commissioning Group (CCG) or practice OR patients identified through social media who have a long-term health condition and/or are taking any medication that requires them to have regular blood tests and have had a medication review in the past six month will be invited to take part in an interview or focus group.
- Public and patient representatives: For the consolidated learning exercise - patient and public representatives who have an understanding of the related medicines management issues in primary care will be invited to take part in an interview or workshop.

SUMMARY:
This study aims to evaluate two interventions designed to make medication prescribing safer, OptimiseRx and PINCER, which are being used in general practices across England. The findings from the evaluation will be used to generate recommendations as to how these interventions can be used sustainably in the long-term.

DETAILED DESCRIPTION:
This study has been designed to evaluate and gain an understanding of the 'real world' implementation, fidelity and medium and longer-term embedding and sustainability of two prescribing safety interventions: the computerised decision support (CDS) tool - Optimize Rx, and PINCER (pharmacist-led information technology intervention for reducing clinically important errors in medication management). The longitudinal process evaluation will involve observations, interviews, focus groups and questionnaires. The consolidated learning exercise, which aims to inform long-term, sustainable intervention use will involve a documentary analysis, interviews, focus groups, development workshops and a synthesis of the evaluation results.

ELIGIBILITY:
Inclusion Criteria:

Staff and stakeholders

* Able to give written informed consent
* 18 years of age or over (no maximum age limit)
* Staff members working in/for a practice or a CCG or the software developer which has received the intervention/s and have direct contact with it/them
* Staff from relevant AHSNs, NHS England, the University of Nottingham or PRIMIS and other relevant staff who have had involvement in the PINCER rollout
* Staff who have either had direct contact with, have an understanding of and/or are in a position to influence wider adoption of the PINCER and OptimseRx interventions (e.g. contracting, IT systems engineer, commissioner, etc.)

Patients

* Able to give written informed consent
* 18 years of age or over (no maximum age limit)
* Patients registered with a general practice who have attended a consultation (or other related activity) for the PINCER intervention, or selected by their clinical care team, or attached to a patient group within a CCG or practice or those identified via social media who are living with a long-term health condition and/or who require regular blood tests to monitor their medication and have had a medication review within the past six months

Members of the public and patient representatives

* Able to give written informed consent
* 18 years of age or over (no maximum age limit)
* Those who have either had direct contact with the PINCER intervention or have an understanding of the related medicines management issues in primary care

Exclusion Criteria:

Staff and stakeholders

* Unable to give written informed consent
* Under 18 years of age

Patients

* Unable to give written informed consent
* Under 18 years of age
* Those considered by their healthcare professional to be inappropriate to recruit due to psycho-social reasons or significant health reasons, e.g. terminal illness/diagnosis.

Members of the public and patient representatives

* Unable to give written informed consent
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Staff and stakeholders will be identified using existing networks and contact details of practice managers, lead GPs, CCG leads, AHSN staff and key stakeholders that are held by the research team. Patients will either be identified by practice staff or through a short, targeted advertisement placed on social media. Public and patient representatives will be identified through healthcare-related patient/public interests groups (e.g. charities, practice group, PPI networks).
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2018-02-16 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary Objective 1. Impact of influential factors in translation, implementation and sustained use of the OptimiseRx and PINCER interventions in the short-term, medium-term or long-term. | Time periods are classified as short-term (< 6 months), medium-term (6-18 months) or long-term (≥ 18 months) implementation
  Semi-structured interviews, focus groups and a questionnaire survey will be conducted to evaluate the contextual factors that influence the nature and extent of translation, implementation and sustained use of the PINCER intervention and prescribing safety indicator (PSI) functions, in particular, across different Academic Health Science Networks (AHSNs) and CCGs over prolonged time periods.
Primary Objective 2. Fidelity of the PINCER intervention delivery and variations in success over time. | Time periods are classified as short-term (< 6 months), medium-term (6-18 months) or long-term (≥ 18 months) implementation
  Semi-structured interviews, focus groups and a questionnaire survey will be conducted to evaluate how the PINCER intervention has been delivered, experienced and has evolved over time in diverse contexts to achieve different degrees of success with particular reference to PSIs.

SECONDARY OUTCOMES:
Secondary Objective 1. Impact and sustained delivery of the PINCER intervention and potential complementary use of OptimseRx and PINCER. | Short-term (< 6 months), medium-term (6-18 months) or long-term (≥ 18 months) implementation
  A documentary analysis, workshops and data synthesis will be conducted to synthesise findings from the primary objectives and from the wider PRoTeCT study along with relevant policies and the perspectives of key stakeholders to generate recommendations for optimal nationwide implementation/impact and sustainable delivery of the OptimiseRx and PINCER interventions which are tailored to different audiences.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Avery, MB, ChB, Principal Investigator — University of Nottingham
Locations (3):
- United Kingdom (3):
  - University of Edinburgh, Edinburgh
  - University of Manchester, Manchester
  - University of Nottingham, Nottingham

IPD SHARING:
Plan to Share IPD: No
Individual patient data will only be shared amongst members of the research team.

REFERENCES:
- [Background] Avery AJ, Rodgers S, Cantrill JA, Armstrong S, Cresswell K, Eden M, Elliott RA, Howard R, Kendrick D, Morris CJ, Prescott RJ, Swanwick G, Franklin M, Putman K, Boyd M, Sheikh A. A pharmacist-led information technology intervention for medication errors (PINCER): a multicentre, cluster randomised, controlled trial and cost-effectiveness analysis. Lancet. 2012 Apr 7;379(9823):1310-9. doi: 10.1016/S0140-6736(11)61817-5. Epub 2012 Feb 21. PMID 22357106
- See also: Medicine Safety and Effective Healthcare Research - PRoTeCT Study Work Package 4 — https://www.nottingham.ac.uk/research/groups/medicinesafetyeffectivehealthcare/protect-study/wp4.aspx